CLINICAL TRIAL: NCT04589598
Title: Comparison Between Femoral Neck System and Multiple Cannulated Screws in Non-displaced Femoral Neck Fracture
Brief Title: Femoral Neck System and Multiple Cannulated Screws in Femoral Neck Fracture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Young-Kyun Lee, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNS-MCS
Record Dates: First submitted 2020-09-27; First posted 2020-10-19 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Femoral Neck Fractures
Keywords: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FNS (Experimental): those who are treated with femoral neck system (FNS)
  Interventions: Device: Femoral Neck System
- MCS (Active Comparator): those who are treated with multiple cannulated screw (MCS)
  Interventions: Device: Multiple Cannulated Screw

INTERVENTIONS:
Device: Femoral Neck System — femoral neck system using bolt and antirotation screw with one/two hole plate
  Arms: FNS
Device: Multiple Cannulated Screw — multiple cannulated screw using 3 or 4 cannulated screw
  Arms: MCS

SUMMARY:
Investigators will compare the clinical outcomes of femoral neck system with conventional multiple cannulated screw in non-displaced femoral neck fracture.

DETAILED DESCRIPTION:
Clinical outcomes include reoperation, loss of fixation, and change of mobility.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* non-displaced femoral neck fracture
* community ambulator

Exclusion Criteria:

* younger than 18 years
* displaced femoral neck fracture
* intertrochanteric fracture
* subtrochanteric fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Reoperation | 3 months
  rate of reoperation
Reoperation | 6 months
  rate of reoperation
Reoperation | 9 months
  rate of reoperation
Reoperation | 12 months
  rate of reoperation
Reoperation | 24 months
  rate of reoperation

SECONDARY OUTCOMES:
loss of fixation | 3 months
  Rate of loss of fixation
loss of fixation | 6 months
  Rate of loss of fixation
loss of fixation | 9 months
  Rate of loss of fixation
loss of fixation | 12 months
  Rate of loss of fixation
loss of fixation | 24 months
  Rate of loss of fixation

OTHER OUTCOMES:
mobility change | 3 months
  Change of mobility
  1. independent community ambulatory
  2. community ambulatory with cane
  3. community ambulatory with crutch, walker
  4. independent household ambulatory
  5. household ambulatory with cane
  6. household ambulatory with crutch, walker
  7. nonfunctional ambulatory
mobility change | 6 months
  Change of mobility
  1. independent community ambulatory
  2. community ambulatory with cane
  3. community ambulatory with crutch, walker
  4. independent household ambulatory
  5. household ambulatory with cane
  6. household ambulatory with crutch, walker
  7. nonfunctional ambulatory
mobility change | 9 months
  Change of mobility
  1. independent community ambulatory
  2. community ambulatory with cane
  3. community ambulatory with crutch, walker
  4. independent household ambulatory
  5. household ambulatory with cane
  6. household ambulatory with crutch, walker
  7. nonfunctional ambulatory
mobility change | 12 months
  Change of mobility
  1. independent community ambulatory
  2. community ambulatory with cane
  3. community ambulatory with crutch, walker
  4. independent household ambulatory
  5. household ambulatory with cane
  6. household ambulatory with crutch, walker
  7. nonfunctional ambulatory
mobility change | 24 months
  Change of mobility
  1. independent community ambulatory
  2. community ambulatory with cane
  3. community ambulatory with crutch, walker
  4. independent household ambulatory
  5. household ambulatory with cane
  6. household ambulatory with crutch, walker
  7. nonfunctional ambulatory

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kyun Lee, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No